CLINICAL TRIAL: NCT05234814
Title: Clinical Study of Auricular Point Seed Burying Combined With Fire Dragon Pot Moxibustion in Perimenopausal Women With Insomnia
Brief Title: Fire Dragon Pot Moxibustion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weihua Yu (Other)
Responsible Party: Sponsor-Investigator, Weihua Yu, Director of nursing department, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-041-01
Record Dates: First submitted 2022-01-28; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Insomnia; Perimenopause
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants with perimenopausal insomnia were randomly divided into a control group and an observation group. Participants in the control group were treated with the traditional Chinese medicine nursing intervention of burying seeds at auricular points. And participants in the observation group were additionally treated with fire dragon pot moxibustion.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group was given the Traditional Chinese Medicine auricular acupuncture point buried seeds therapy.
  Interventions: Other: Traditional Chinese Medicine auricular acupuncture point buried seeds therapy
- Observation group (Experimental): The observation group was given the auricular acupuncture point buried seeds therapy plus the fire dragon pot moxibustion therapy.
  Interventions: Other: Traditional Chinese Medicine auricular acupuncture point buried seeds therapy plus the fire dragon pot moxibustion therapy.

INTERVENTIONS:
Other: Traditional Chinese Medicine auricular acupuncture point buried seeds therapy plus the fire dragon pot moxibustion therapy. — Fire dragon pot moxibustion treatment The main acupuncture points are as follows: Fengchi, Jianjin, Dazhui, Feiyu, Xinyu, Ganyu, Piyu, Shenyu, etc (all acupuncture points are positioned according to the national standard: GB/T12346-2006).
  Ear acupuncture seed burial method According to "Ear Acupuncture Therapy" [6], the main acupuncture points were Shenmen, subcortical, sympathetic, endocrine, kidney, heart, liver and spleen (all acupuncture points were positioned according to the national standard: GB/T12346-2006).
  Arms: Observation group
Other: Traditional Chinese Medicine auricular acupuncture point buried seeds therapy — Ear acupuncture seed burial method According to "Ear Acupuncture Therapy" [6], the main acupuncture points were Shenmen, subcortical, sympathetic, endocrine, kidney, heart, liver and spleen (all acupuncture points were positioned according to the national standard: GB/T12346-2006).
  Arms: Control group

SUMMARY:
Insomnia in perimenopausal women is normal. Studies have shown that insomnia occurs in 75-81% of perimenopausal women and is 2.4 times more common than in premenopausal participants. Western medicine often uses sedative sleeping drugs in the treatment of insomnia in perimenopausal women, which have better effects but have more side effects, and whether they are suitable for long-term application is still controversial. Non-pharmacological traditional therapies in Traditional Chinese Medicine have achieved significant clinical efficacy in the treatment of perimenopausal insomnia patients in recent years. This study aims to explore the efficacy of auricular point seed burying combined with fire dragon pot moxibustion in the treatment of the insomnia symptoms of perimenopausal women.

DETAILED DESCRIPTION:
Female menopausal participants often experience physical and psychological symptoms such as anxiety, depression and sleep disturbances due to the weakening of the ovaries and hormonal changes in the body, with insomnia being the most typical symptom. Studies have shown that insomnia occurs in 75-81% of perimenopausal women and is 2.4 times more common than in premenopausal participants. The main symptoms are difficulty falling asleep, early awakening and easy waking, which may be accompanied by anxiety, irritability and sweating. Long-term insomnia will lead to impairment of multi-system function and endanger the physical and mental health of perimenopausal women. The treatment of insomnia during menopause in Western medicine is mainly based on pharmacological treatment, but it is controversial whether it is suitable for long-term clinical application due to drug dependency and other side effects. Non-pharmacological traditional therapy in Traditional Chinese Medicine is more acceptable to participants because of its efficacy, non-chemical and non-toxic side effects. Furthermore, it has been used in the clinical application of insomnia in perimenopausal participants with good efficacy in recent years. In this study, we used auricular seeds burying combined with fire dragon pot moxibustion as an appropriate Chinese medicine technique to treat perimenopausal women with insomnia, hoping to improve the life quality of perimenopausal women with insomnia.

ELIGIBILITY:
Inclusion Criteria:

* All participants met the diagnosis of perimenopausal insomnia as described in the Chinese Guidelines for the Diagnosis and Treatment of Adult Insomnia (2017 Edition).
* Pittsburgh Sleep Quality Index (PSQI) >7.
* Insomnia at least 3 times per week and lasting for more than 1 month.
* Onset around menopause with menstrual disorders.
* No contraindications to auricular seed burial and fire dragon pot moxibustion treatment
* Informed consent.

Exclusion Criteria:

* Those with a duration of less than 1 week or those who have received other relevant treatment within the last month that affects the observation of efficacy
* Secondary insomnia due to physical illness or psychological disorders.
* Participants with severe co-morbidities and psychiatric disorders.
* Those who refuse to cooperate with treatment.
* Those who use other methods of treatment during the treatment period, which affects the judgment of efficacy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The score of Pittsburgh Sleepiness Quantifier Inventory | one month
  The score of Pittsburgh Sleepiness Quantifier Inventory (PSQI) was compared between the two groups of patients before and after the intervention (For details, please refer to the literature: The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research). A PSQI score <7 is considered good sleep quantity and ≥7 is poor sleep quality, and the higher the patient score, the worse the sleep quality.

SECONDARY OUTCOMES:
Adverse reactions | one month
  Observe whether erythema, blisters, allergic and other adverse reactions are appearing

CONTACTS AND LOCATIONS:
Overall Officials: Weihua Yu, Dr., Principal Investigator — The Third Affiliated Hospital of Anhui Medical University
Locations (1):
- The Third Affiliated Hospital of Anhui Medical University (The first people ' s Hospital of Hefei), Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
The data is available upon reasonable request